CLINICAL TRIAL: NCT05637645
Title: Different Approaches of Spinal Anesthesia in Patients Undergoing Cesarean Section: Midline, Paramedian and Taylors Approach
Brief Title: Different Approaches of Spinal Anesthesia in Patients Undergoing Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bahawal Victoria Hospital Bahawalpur (Other)
Responsible Party: Principal Investigator, Muhammad Ali Fayyaz, Dr Muhammad Ali Fayyaz, Bahawal Victoria Hospital Bahawalpur
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 1229/DME/QAMC Bahawalpur
Record Dates: First submitted 2022-11-21; First posted 2022-12-05 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Post-Dural Puncture Headache; Hypotension; Spinal Shock; Hematoma; Bradycardia; Meningitis; Respiratory Failure
Keywords: Midline approach; Spinal anesthesia; cesarean section; Taylors approach
MeSH Terms: conditions — Post-Dural Puncture Headache; Hypotension; Hematoma; Bradycardia; Meningitis; Respiratory Insufficiency | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants are assigned to three groups in parallel for the duration of the study Group M for participants are given spinal anesthesia through Midline approach Group P for participants are given spinal anesthesia through Paramedian approach Group T for participants are given spinal anesthesia through Taylors approach
Who Masked: Participant, Care Provider
Masking Description: Health care workers including nurses paramedical staff and ward boys may be masked from this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group M (Active Comparator): It will involve participants who are given spinal anesthesia through midline approach.
  Interventions: Procedure: Midline Approach
- Group P (Active Comparator): It will involve participants who are given spinal anesthesia through paramedian approach.
  Interventions: Procedure: Paramedian Approach
- Group T (Active Comparator): It will involve participants who are given spinal anesthesia through Taylors approach.
  Interventions: Procedure: Taylors approach

INTERVENTIONS:
Procedure: Midline Approach — In the midline approach, the spinal approach to the intrathecal space is midline with a straight line shot. After infiltration with lidocaine, the spinal needle is introduced into the skin, angled slightly cephalic. The needle traverses the skin, followed by subcutaneous fat. A single dose of 12.5mg of 0.5% bupivacaine (preservative free) will be used for the spinal anesthetic, the effects of this will last approximately 2 hours.
  Other Names: Spinal needle; Bupivacaine
  Arms: Group M
Procedure: Paramedian Approach — The paramedian approach involves inserting the spinal needle 1 cm away from the midline in medial direction. A single dose of 12.5mg of 0.5% bupivacaine (preservative free) will be used for the spinal anesthetic, the effects of this will last approximately 2 hours.
  Other Names: Spinal needle; Bupivacaine
  Arms: Group P
Procedure: Taylors approach — his arm will have the procedure of spinal anesthetic performed via 'Taylor's approach' which is a paramedian approach to interspace L5 - S1. A single dose of 12.5mg of 0.5% bupivacaine (preservative free) will be used for the spinal anesthetic, the effects of this will last approximately 2 hours.
  Other Names: Spinal needle; Bupivacaine
  Arms: Group T

SUMMARY:
The goal of this clinical trial is to compare different approaches of spinal anesthesia in pregnant females who are having cesarean section. The main aim is

• Which approach is better in terms of avoiding intraoperative and post operative complications

Participants will be given anesthesia by

1. Midline approach
2. paramedian approach
3. Taylors approach

DETAILED DESCRIPTION:
1. Introduction to study:

   Different techniques and modalities are used to anesthetize the patient for the smooth conduction of surgery including, general anesthesia, spinal anesthesia, different types of regional anesthesia and monitored anesthesia care.1 According to the authors' knowledge, limited local studies are available that compare midline to the paramedian approach, Taylor's approach and Transforaminal approach of spinal anesthesia in the context of occurrence of post-dural puncture headaches, backache, hematoma, paresthesia, pulse, blood pressure, respiratory rate, temperature and urine output.3
2. Problem statement:

   Post-dural puncture headache is defined as a bilateral headache that develops within 7 days after dural puncture. It characteristically worsens 15 minutes after resuming sitting position and improves or disappears within 30 minutes of resuming supine position. It can be managed with medical as well as autologous epidural blood patch. It may result in prolonged recovery and delayed mobilization as well as psychosomatic side effects. More sinister side effects like subdural hematoma and seizures are rare but may prove fatal.2 The exact mechanism of development of postdural puncture headache is unclear. The postulated pathogenesis involves cerebrospinal fluid (CSF) leak through the dural puncture site resulting in intracranial hypotension leading to traction on intracranial structures and vasodilatation of cerebral vessels resulting in headache.2
3. Objectives of this research:

   i) To find out frequency of Post-dural puncture headache (PDPH) in patients with different groups undergoing different approaches of spinal anesthesia.

   ii) Impact of different approaches of spinal anesthesia on complications of spinal anesthesia. Complications are related to either exaggerated physiologic responses or needle/catheter insertion and include:
   * Post-dural-puncture headache (PDPH)
   * Hypotension and bradycardia secondary to sympathetic blockade
   * Hypothermia
   * Respiratory failure resulting from a "high spinal/block"
   * Urinary retention
   * Spinal infection, including aseptic meningitis
   * Spinal or epidural hematoma
   * Nerve or spinal cord damage, possibly resulting in paralysis
   * Pain iii) Impact of different approaches of spinal anesthesia on vitals (pulse, BP, temperature, respiratory rate, spO2 and urine output) intraoperatively and postoperatively.
4. Limitation of the study:

   The study will be limited to patients undergoing cesarean section. No general population will be involved.
5. Methodology Paper based questionnaire will be filled out by doctors on duty during pre-operative, operative and post operative period of patients. The study will be a comparative study based on CONSORT randomized control trial in which different groups based on approaches i.e. midline, paramedian, Taylor's and transforaminal approach, will be made. Sampling will involve lottery method. Data will be analyzed by IBM SPSS Statistics Digital Software version 20.0. Data analysis will be done by comparing different groups based on approaches i.e. midline, paramedian, Taylor's and transforaminal approach.

Exclusion Criteria

1. Patients who refuse to participate in study.
2. More than 3 attempts of lumber puncture
3. Previously having migraines of PDPH
4. Hb less than 7
5. INR more than 1.2
6. Previous C-section more than 5
7. Patients with placenta previa, accrete, percreta and increta
8. NPO less than 6 hours preoperatively
9. Patients from gynecological department other than C-section

Study Setting:

Emergency Operation Theatre, Bahawal Victoria Hospital, Bahawlpur.

6. Ethical Consideration Points:

1. Applied for ERC approval at DME QMC.
2. Obtained written consent from study participants.
3. Given autonomy to study participants.
4. Maintained confidentiality of the data obtained.
5. Given some beneficial effects to study participants.
6. No harm to study participants.
7. Non-maleficence.
8. Justice and fair play.
9. No conflict of interest among study authors.
10. Study funding source mentioned if received from outside, other than study authors.
11. Appropriate treatment availability at our institution for diseased subjects.
12. In case of any referral, arrangements for it would be done.
13. Study results dissemination to study participants would be done.
14. Plagiarism check report within appreciate limits (less than 20%) is checked by given HEC licensed criteria.
15. Contribution of each author made in conducting the study is mentioned with his/her name, proper designation and contact number/email.

ELIGIBILITY:
Exclusion Criteria:

1. Patients who refuse to participate in study.
2. More than 3 attempts of lumber puncture
3. Previously having migraines of PDPH
4. Hb less than 7
5. INR more than 1.2
6. Previous C-section more than 5
7. Patients with placenta previa, accrete, percreta and increta
8. NPO less than 6 hours preoperatively
9. Patients from gynecological department other than C-section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Post-dural-puncture headache (PDPH) | 1 month
  PDPH is the most common complication after spinal anesthesia. Our study is based on prevention of PDPH using different approach in spinal anesthesia

SECONDARY OUTCOMES:
Hypotension and bradycardia secondary to sympathetic blockade | 1 day
Hypothermia | 1 day
Respiratory failure | 5 days
Spinal Shock | 1 day
Urinary retention | 1 month
Meningitis | 1 month
Hematoma | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ali Fayyaz, MBBS, BSC, Principal Investigator — Bahawal Victoria Hospital Bahawalpur
Locations (4):
- Pakistan (4):
  - Bahawal Victoria Hospital Bahawalpur, Bahawalpur, Punjab Province
  - Bahawalpur Medical & Dental College Bahawalpur, Bahawalpur, Punjab Province
  - Hameed Latif Hospital, Lahore, Punjab Province
  - Laeeque Rafiq Hospital (LRH) Multan, Multan, Punjab Province

IPD SHARING:
Plan to Share IPD: No
This clinical trial is going to be publish in an international journal. To prevent the data from being available to every researcher will not make any difference.

REFERENCES:
- [Result] Hempel V. [Spinal anesthesia for cesarean section]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2001 Jan;36(1):57-60. doi: 10.1055/s-2001-10239-8. German. PMID 11227314
- [Result] Buddeberg BS, Bandschapp O, Girard T. Post-dural puncture headache. Minerva Anestesiol. 2019 May;85(5):543-553. doi: 10.23736/S0375-9393.18.13331-1. Epub 2019 Jan 4. PMID 30621376
- [Result] Fernandes NL, Dyer RA. Anesthesia for Urgent Cesarean Section. Clin Perinatol. 2019 Dec;46(4):785-799. doi: 10.1016/j.clp.2019.08.010. Epub 2019 Aug 14. PMID 31653308
- [Result] Bernstein K, Hussey H, Hussey P, Gordo K, Landau R. Neuro-anesthesiology in pregnancy. Handb Clin Neurol. 2020;171:193-204. doi: 10.1016/B978-0-444-64239-4.00010-2. PMID 32736750
- [Result] Parikh KS, Seetharamaiah S. Approach to failed spinal anaesthesia for caesarean section. Indian J Anaesth. 2018 Sep;62(9):691-697. doi: 10.4103/ija.IJA_457_18. PMID 30237594

DOCUMENTS (1):
  • Informed Consent Form (2022-11-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT05637645/ICF_000.pdf